CLINICAL TRIAL: NCT06282029
Title: Acceptance and Commitment Therapy-based Group Therapy for Mental Health After Stroke - a Pilot Study
Brief Title: ACT-group for Stroke Survivors (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Collaborators: Bielefeld Young Researchers' Fund (Unknown)
Responsible Party: Principal Investigator, Simon Ladwig, Principal Investigator, Bielefeld University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I-2720-0018-0003
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Intracerebral Hemorrhage; Depressive Symptoms; Anxiety; Stress
Keywords: Acceptance and Commitment Therapy; Group therapy; Pilot study; Feasibility
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Depression; Anxiety Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: This pilot study includes a pre-/post test of a small intervention sample without control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Group therapy
  Interventions: Behavioral: Group Therapy

INTERVENTIONS:
Behavioral: Group Therapy — Acceptance and Commitment Therapy based group therapy

SUMMARY:
The goal of this clinical pilot trial is to test the feasibility, acceptance and preliminary efficacy of an adapted group psychotherapy manual in stroke survivors with psychological stress. The main questions it aims to answer are:

* Is the group therapy feasible?
* Is the group therapy accepted by stroke survivors and therapists?
* Are there first indications on the efficacy of the group therapy to improve mental health?

Participants will take part in 8 weekly group therapy sessions of 90 minutes each.

DETAILED DESCRIPTION:
This trail aims to investigate the feasibility, acceptance and preliminary efficacy of a group therapy manual based on Acceptance and Commitment Therapy. The manual is an adaptation of "Living Well with Neurological Conditions" (Hill et al., 2017), which was conducted in groups with acquired brain injury in general. The manual was translated to German and adapted to the needs of stroke survivors who are often older, have more comorbidities and specific neurological impairments. Session length was reduced from 165 minutes to 90 minutes. The program includes 8 weekly sessions. In addition, outcome questionnaires were translated to German and all measures are translated into plain language to increase accessibility.

ELIGIBILITY:
Inclusion Criteria:

* Value above a cut-off on one of the DASS-21 subscales (depression > 10, anxiety > 6, and stress > 10)
* Sufficient cognition and language ability (clinical rating)
* Sufficient therapy motivation (clinical rating)

Exclusion Criteria:

* Behavioral disorders (e.g., high irritability or apathy in clinical rating)
* Other severe mental disorder (dementia, psychosis, personality disorders, intellectual disability)
* Parallel psychotherapy or neuropsychological therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Drop-out rate | Until end of last session, presumably 8 weeks
  Rate of participants discontinuing the group therapy ≤ 20% in each group. Drop-out rate is one indicator of feasibility.
Session adherence | Until end of last session, presumably 8 weeks
  Mean rate of participants attending sessions ≥ 80% in each group. Attendance is assessed each session and averaged over all 8 sessions. Session adherence is one indicator of feasibility.
Homework completion | Until end of last session, presumably 8 weeks
  Mean rate of participants completing homework ≥ 50% in each group. Mean rate of participants attending sessions ≥ 80% in each group. Homework completion is assessed each session and averaged over all 8 sessions. Homework completion is one indicator of feasibility.
Completion of outcome measures | Before first and after last session (time frame = 8 weeks)
  Mean rate of completed outcome measures ≥ 80% in each group. Rate is calculated based on number of completed items in all questionnaires. Completion of outcome measures is one indicator of feasibility.
Treatment fidelity | Until end of last session, presumably 8 weeks
  Treatment fidelity ≥ 80% in each group. Two randomly selected sessions are video-recorded. A research assistant then applies self-developed checklists for the respective sessions to assess if therapists adhere to manual instructions and contents. Treatment fidelity is one indicator of feasibility.
Group therapy session questionnaire - patients (Zoubek, 2013; Plain German) | Until end of last session, presumably 8 weeks
  Patients rate acceptance for each session and the whole group therapy.
Group therapy session questionnaire - therapists (Zoubek, 2013; Plain German) | Until end of last session, presumably 8 weeks
  Therapists rate acceptance for each session and the whole group therapy.
Acceptance and Action Questionnaire-Acquired Brain Injury (Sylvester, 2011; Plain German) | Before first and after last session, presumably 8 weeks
  Measure of psychological flexibility to investigate efficacy. Scores range from 0 to 36 with higher values indicating higher inflexibility.
Depression and Anxiety Stress Scales-21 (Lovibond, 1995; Plain German) | Before first and after last session, presumably 8 weeks
  Measure of psychological burden to investigate efficacy. Scores range from 0 to 63 with higher values indicating higher burden.

SECONDARY OUTCOMES:
Valuing Questionnaire (Smout, 2014; Plain German) | Before first and after last session, presumably 8 weeks
  Measure of valued living to investigate efficacy. Scores range from 0 to 60 with higher values indicating higher value-congruent living.
Self-as-context scale (Zettle, 2018; Plain German) | Before first and after last session, presumably 8 weeks
  Measure of self as context to investigate efficacy. Scores range from 10 to 70 with higher values indicating a perspective closer to self-as-context.
Patient Health Questionnaire-9 (Kroenke, 2001; Plain German) | Before first and after last session, presumably 8 weeks
  Measure of depressive symptoms to investigate efficacy. Scores range from 0 to 27 with higher values indicating more severe depressive symptoms.
Generalized Anxiety Disorder-7 (Spitzer, 2006; Plain German) | Before first and after last session, presumably 8 weeks
  Measure of anxiety symptoms to investigate efficacy. Scores range from 0 to 21 with higher values indicating more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Ladwig, PhD, Principal Investigator — Bielefeld University
Locations (1):
- University Neuropsychological Outpatient Clinic, Bielefeld, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill G, Hynd N, Price J, Evan S, Moffitt J, Brechin D. Living well with neurological conditions. South Tees Hospitals NHS Fundation Trust. 2017.
- [Background] Zoubek, K. (2013). Prozessevaluation einer kognitiv-verhaltenstherapeutischen Gruppentherapie bei Diabetes und Depression: Entwicklung und Validierung der Patienten- und Therapeuten-Gruppentherapiestundenbögen (GTS-P, GTS-T, GTS-TP) zur Vorhersage des Therapieerfolgs. [Dissertation, Johannes Gutenberg-Universität Mainz]. OpenScience JGU Mainz.
- [Background] Sylvester, M. (2011). Acceptance and Commitment Therapy for improving adaptive functioning in persons with a history of pediatric acquired brain injury. [Doctoral dissertation, University of Nevada]. ProQuest
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Smout, M., Davies, M., Burns, N., & Christie, A. (2014). Development of the valuing questionnaire (VQ). Journal of Contextual Behavioral Science, 3(3), 164-172.
- [Background] Zettle, R. D., Gird, S. R., Webster, B. K., Carrasquillo-Richardson, N., Swails, J. A., & Burdsal,C. A. (2018). The Self-as-Context Scale: Development and preliminary psychometric properties. Journal of Contextual Behavioral Science, 10, 64-74
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT06282029/Prot_SAP_000.pdf